CLINICAL TRIAL: NCT02318758
Title: Randomized, Single Dose, 4-Way Cross-over Study to Investigate the Pharmacokinetic Interaction of Oral Treprostinil and Ethanol in Healthy Volunteers
Brief Title: Pharmacokinetic Interaction of Oral Treprostinil and Ethanol in Healthy Volunteers
Acronym: TDE-PH-125
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: TDE-PH-125
Record Dates: First submitted 2014-09-15; First posted 2014-12-17 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: This is a healthy volunteer study.
MeSH Terms: interventions — treprostinil; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Comparison 1 (Active Comparator): UT-15C 1 mg alone
  Interventions: Drug: UT-15C
- Comparison 2 (Active Comparator): UT-15C 1 mg plus ethanol (simultaneously)
  Interventions: Drug: UT-15C; Other: ethanol
- Comparison 3 (Active Comparator): UT-15C 1 mg administered 1 hour before ethanol
  Interventions: Drug: UT-15C; Other: ethanol
- Comparison 4 (Active Comparator): UT-15C 1 mg administered 1 hour after ethanol
  Interventions: Drug: UT-15C; Other: ethanol

INTERVENTIONS:
Drug: UT-15C — sustained release oral treprostinil
  Other Names: Oral treprostinil
Other: ethanol — Absolut 100 vodka
  Other Names: alcohol
  Arms: Comparison 2; Comparison 3; Comparison 4

SUMMARY:
A study to assess the interaction of acohol and oral treprostinil.

DETAILED DESCRIPTION:
This study will compare the effects of ethanol on the PKs of a 1 mg dose of UT-15C in healthy volunteers to determine the in vivo effects of ethanol, including the timing of ethanol consumption in relation to UT-15C ingestion.

This is an open-label, randomized, single-center, four-way (period), crossover study in which 28 healthy volunteers will receive a single 1 mg oral dose of UT-15C and/or ethanol. Eligible subjects will be randomly assigned to one of four treatment sequences such that all subjects will receive all four sequences in a pre-specified order.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily gives informed consent to participate in the study.
2. Women of child bearing potential includes any female who has experienced menarche and who has not undergone successful surgical sterilization. Women of childbearing potential must practice true abstinence from intercourse when it is in line with their preferred and usual lifestyle, or use two different forms of highly effective contraception for the duration of the study, and for at least 30 days after discontinuing study medication. Medically acceptable forms of effective contraception include: (1) approved hormonal contraceptives (such as birth control pills), (2) barrier methods used with a spermicide, (3) an intrauterine device, or (4) partner vasectomy. For women of childbearing potential, a negative urine pregnancy test is required at Screening and Baseline prior to initiating study medication.
3. The subject, if male, must use a condom during the length of the study, and for at least 48 hours after discontinuing study medication.
4. Healthy male and female subjects aged 21-55 years of age at the time of signing the informed consent.
5. Weight between 55 and 100 kg, with a BMI between 19.0-29.9 kg/m2, inclusive for female subjects and weight between 55 and 120 kg, with a BMI between 19.0-32.0 kg/m2, inclusive for male subjects.
6. Regular consumption of ethanol with no recent changes in pattern of consumption
7. In the opinion of the Principal Investigator, the subject is able to communicate effectively with study personnel, and is considered reliable, willing and likely to be cooperative with protocol requirements, including attending all study visits.

Exclusion Criteria:

1. The subject is pregnant or lactating.
2. Subject has any clinically relevant abnormality identified during the screening physical examination, 12-lead ECG, or laboratory examinations.
3. Subject has a history of anaphylaxis, a previous documented hypersensitivity reaction, or a clinically significant idiosyncratic reaction to any drug.
4. Subject has a clinically significant history of neurological, cardiovascular, respiratory, endocrine, hematological, hepatic, renal, gastrointestinal, genitourinary, pulmonary, and/or musculoskeletal disease; glaucoma; a psychiatric disorder, or any other chronic disease, whether controlled by medication or not.
5. Subject has a history of postural hypotension, or unexplained syncope.
6. Subject has a blood pressure that is less than 85 mmHg systolic or 50 mmHg diastolic at Screening or Baseline.
7. Subject has a pulse rate that is greater than 90 bpm after sitting at rest for 5 minutes at Screening or Baseline.
8. Subject has a blood pressure that is greater than 150 mmHg systolic or 90 mmHg diastolic at Screening or Baseline.
9. Subject has a predisposing condition that could interfere with the absorption, distribution, metabolism, or excretion of drugs.
10. Subject has tested positive at the screening visit for HIV infection, HBsAg, or the HCV antibody.
11. Subject currently uses tobacco products or has a history of tobacco use within two months prior to Baseline.
12. Subject has a history of ethanol abuse or a history of or current impairment of organ function reasonably related to ethanol abuse.
13. Subject has a history of or current evidence of abuse of licit or illicit drugs, including a positive urine screen for drugs of abuse at Screening or Baseline.
14. Subject has a history of abnormal bleeding tendencies.
15. Subject has donated blood or plasma or has lost a significant volume of blood within four weeks prior to Baseline.
16. Subject has clinically significant abnormal laboratory values in the opinion of the treating Investigator.
17. Subject has participated in a research study within the last 30 days.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of oral treprostinil (Cmax) | Subjects will be enrolled for 24 days

SECONDARY OUTCOMES:
Safety and tolerability via laboratory values, collection of adverse events, vital signs and electrocardiogram. | Subjects will be enrolled for 24 days

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Laurent, MD, Principal Investigator — PPD Development, LP
Locations (1):
- PPD International, Austin, Texas, United States